CLINICAL TRIAL: NCT02246049
Title: A Multicenter, Clinical Phase II Study of FOLFOXIRI With Bevacizumab As First-line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: A Multicenter, Clinical Study of FOLFOXIRI With Bevacizumab As First-line Therapy in Patients With mCRC
Acronym: QUATTRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EPS Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUATTRO
Record Dates: First submitted 2014-09-12; First posted 2014-09-22 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
Keywords: Metastatic colorectal cancer, bevacizumab, FOLFOXIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOXIRI plus bevacizumab (Experimental): Induction therapy is followed by the maintenance therapy.
  [Induction treatment:FOLFOXIRI plus bevacizumab] Administered for a maximum of 12 cycles. BV: 5mg/kg (d.i.v.) L-OHP: 85 mg/sq.m (d.i.v.) CPT-11:165mg/sq.m (d.i.v.) l-LV:200mg/sq.m (d.i.v.) 5-FU:3,200mg/sq.m (c.i.v.) Administered every 2 weeks.
  [Maintenance treatment:5-FU / I-LV plus bevacizumab] BV:5mg/kg (d.i.v.) l-LV:200mg/sq.m (d.i.v.) 5-FU:3,200mg/sq.m (c.i.v.) Administered every 2 weeks.
  Interventions: Biological: Bevacizumab; Drug: 5-fluorouracil; Drug: Irinotecan hydrochloride; Drug: Leucovorin calcium; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: BV
Drug: 5-fluorouracil — Given IV
  Other Names: 5-FU
Drug: Irinotecan hydrochloride — Given IV
  Other Names: CPT-11
Drug: Leucovorin calcium — Given IV
  Other Names: I-LV
Drug: Oxaliplatin — Given IV
  Other Names: L-OHP

SUMMARY:
The purpose of this study to assess efficacy and tolerability of combination therapy FOLFOXIRI with Bevacizumab (BV) as a first-line therapy in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a single-arm, multicentre phase II study evaluating the efficacy and safety of Bevacizumab (BV) in combination with oxaliplatin, irinotecan hydrochloride, fluorouracil, and leucovorin calcium regimen ( FOLFOXIRI +BV ; Falcone et al. ASCO2013) as first-line treatment for Japanese metastatic colorectal cancer patients.

This study is composed two steps because of collecting safety issue in Japanese patient.

As First step (Step 1), It assess on the initial safety information in ten Japanese patients of the end of 2nd cycle. it is evaluated by DMC.

In parallel with the confirmation of the initial safety issue, register up to 65 cases in total and Step 1 patient, to evaluate the efficacy and safety (Step2).

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed consent.
2. Histopathologically proven diagnosis of colorectal cancer (adenocarcinoma) excluding vermiform appendix cancer and proctos cancer.
3. Not resectable metastatic colorectal cancer
4. Age at enrollment is >= 20 and <= 75 years
5. ECOG PS < 2 if age < 70 years, ECOG PS = 0 if age = 71-75 years
6. One or more measurable lesion in RECIST ver.1.1 criteria according to contrast enhanced CT chest / abdomen / pelvis diagnosis.
7. Not previously treated with chemotherapy. ( Previous adjuvant by fluoropyrimidine monotherapy is allowed if more than 24 weeks have elapsed between the end of adjuvant therapy and first relapse.)
8. Vital organ functions (listed below) are preserved within 2 weeks prior to entry. Data recorded nearest to the entry should be referred. Blood transfusion or erythropoiesis stimulating agents less than 2 weeks prior to the tests are not allowed.

   Neu. >= 1,500/cubicmillimeter Pt. >= 100,000/cubicmillimeter Hb. >= 9.0 g/dL T-bil. <= upper limit of normal (ULN)*1.5 AST and ALT,ALP <= upper limit of normal (ULN)*2.5 (<= ULN*5 in case of liver metastasis) Serum creatinine <= upper limit of normal (ULN) *1.5 PT-INR < 1.5 Proteinuria <= 2+
9. UGT1A1 genotype tested. Categorized into Wild or single Hetero.

Exclusion Criteria:

1. Previously treated with irradiation to bone marrow constituting 20% or more of irradiation field.
2. Untreated brain metastases or spinal cord compression or primary brain tumors.
3. History of CNS disease.[except for asymptomatic Lacunar stroke]
4. Requiring chronic systemic corticosteroid treatment.
5. Current or recent ongoing treatment with anticoagulants.
6. Clinically significant cardiovascular disease for example cerebrovascular accidents, myocardial infarction, unstable angina, congestive heart failure, serious cardiac arrhythmia requiring medication.
7. Treatment with any investigational drug within 4 weeks.
8. Patient with Uncontrolled hypertension, Uncontrolled diabetes, Uncontrolled diarrhea, >=grade 1 peripheral neuropathy, Active peptic ulcer, Non-healing wound, Clinically important diseases.
9. Major surgical procedure within 28 days prior to study treatment start, open biopsy, or significant traumatic injury, or anticipation of the need for major surgical procedure.[except for implantation of central venous catheter and port system.]
10. Lack of physical integrity of the upper gastrointestinal tract.
11. Pregnant women, lactating woman , positive by pregnancy test , wishing to become pregnant, and Sexually active males.
12. Hepatitis B or hepatitis C. Evidence of HIV infection.
13. Previous Chemotherapy for other organs.
14. Other active co-existing malignancies.
15. History / Presence of thrombosis within 1 year requiring medication.
16. History / Presence of paralytic ileus, obstruction or gastrointestinal perforation.
17. Malignant coelomic fluid required drainage.
18. History of allergy to Chinese hamster ovary cell proteins, or any of the components of the study medications.
19. History of fluoropyrimidine severe side effects caused by DPD defect.
20. Interstitial pneumonitis or pulmonary fibrosis.
21. Evidence or requiring systemic treatment for Infectious disease.
22. Patient who is judged by the investigator to be inappropriate for study participation for any reason.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 10 months | PFS rate at 10 months from study entry
  PFS by investigator-reported measurements according to CT image. PFS was calculated from the day of treatment start to the first observation of progression disease (PD) or death from any cause.
  PD was defined as Overall Response by RECIST criteria v1.1 according to CT image.

SECONDARY OUTCOMES:
Response rate (RR) by central review. | Up to 18 months
  Response evaluation was performed according to RECIST criteria v1.1.
Response rate (RR) by investigator-reported measurements. | Up to 30 months
  Response evaluation was performed according to RECIST criteria v1.1.
PFS by central review according to CT image. | Up to 18 months
  PFS was calculated from the day of treatment start to the first observation of progression disease (PD) or death from any cause.
Overall survival (OS) | Up to 30 months
  OS was calculated from the day of registration in this study to death from any cause.
Efficacy by RAS status ; RR,PFS,OS | Up to 30 months
  RR,PFS,OS according to tumor RAS status.
Incidence of adverse events | Up to 30 months
  Adverse events were evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0. All adverse events was collected in duration from starting treatment to whichever shorter "after 30 days from withdrawal treatment" or "later treatment was started".
Time to treatment-failure | Up to 30 months
Completion rate in Induction treatment | Up to 30 months
Relative Dose Intensity | Up to 30 months
Treatment duration | Up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kato, M.D., Ph.D, Principal Investigator — Department of Surgery, National Hospital Organization Osaka National Hospital.; Akiyoshi Kanazawa, M.D., Ph.D, Principal Investigator — Department of Surgery, Shimane Prefectural Central Hospital.
Locations (1):
- EPS Corporation, Shinjuku, Tokyo, Japan